CLINICAL TRIAL: NCT07395557
Title: The Effects of Education and Counseling Applied Via Mobile Application Based on the Pender Health Promotion Model on Symptom Severity, Quality of Life and Sleep Quality in Women With Urinary Incontinence During Menopause
Brief Title: Effect of a Pender Model-Based Mobile App on Symptom Severity, Quality of Life, and Sleep in Menopausal Women With Urinary Incontinence
Acronym: UI Sleep QoL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Pınar Doğancı, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200902038
Record Dates: First submitted 2025-09-15; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Menopause; Urinary Incontinence; Mobile Applications; Quality of Life; Sleep
Keywords: Menopause; Urinary Incontinence; Mobile Applications; Quality of Life; Sleep; Pender's Health Promotion Model
MeSH Terms: conditions — Urinary Incontinence | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with urinary incontinence receiving mobile-based exercise interventions (Experimental): Being a woman aged between 40 and 65
  Being postmenopausal
  Experiencing urinary incontinence
  Being literate
  Having sufficient proficiency in understanding and speaking Turkish
  Having no diagnosed psychiatric disorders
  Owning a smartphone with Android or iOS operating system and having internet access
  Volunteering to participate in the study
  Interventions: Behavioral: Education and counseling delivered via a mobile application based on Pender's Health Promotion Model
- Individuals receiving routine care (No Intervention): Individuals will receive routine care, and no intervention will be applied.

INTERVENTIONS:
Behavioral: Education and counseling delivered via a mobile application based on Pender's Health Promotion Model — Questionnaires will be given as a pre-test at the initial meeting. After randomization, the intervention group will have a mobile app installed and create a profile. They will read modules, do daily exercises, and fill follow-up forms. Mini-tests after each module require at least 75% correct to continue; otherwise, the module is reread. The intervention lasts 8 weeks, covering fluid intake, urine tracking, diet, healthy eating, bladder, and Kegel exercises. Studies show exercises reduce urinary incontinence after 6 weeks, so 8 weeks is planned. After intervention, questionnaires will be repeated. The control group gets no intervention but completes questionnaires at start and end. Weekly calls support the intervention group's motivation and symptom monitoring; the control group is called at weeks 3 and 8. After the study, the app is given to controls. Data is used only for research and accessible to researchers and admins.
  Arms: Individuals with urinary incontinence receiving mobile-based exercise interventions

SUMMARY:
Objective: This randomized controlled trial aims to examine the effects of education and counseling delivered through a mobile application based on the Pender Health Promotion Model on symptom severity, quality of life, and sleep quality in menopausal women with urinary incontinence.

Methods: The study was conducted at Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, targeting women who presented to the urology outpatient clinic and met the inclusion criteria. The sample consisted of 82 participants, with 41 women in the intervention group and 41 in the control group. To account for potential dropouts during the mobile intervention, the sample size was increased by 20% above the calculated requirement.

Data collection tools included the Descriptive Information Form, Incontinence Quality of Life Questionnaire (I-QOL), Incontinence Severity Index (ISI), International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), and Pittsburgh Sleep Quality Index (PSQI).

The intervention group received an 8-week mobile application-based education program developed in line with the Pender Health Promotion Model. Additionally, participants in the intervention group were contacted twice weekly by phone for counseling and support. The control group received no educational intervention but was assessed with pre-test and post-test measurements.

Results: Data were analyzed using descriptive statistics, independent and paired sample t-tests, one-way and repeated measures ANOVA, Pearson correlation analysis, and chi-square tests for group homogeneity. The study aims to determine whether the mobile application-based intervention significantly improves urinary incontinence symptoms, quality of life, and sleep quality compared to the control group.

Conclusion: This study may provide evidence supporting the use of mobile health interventions based on health promotion models like Pender's to enhance the management and overall well-being of menopausal women with urinary incontinence.

DETAILED DESCRIPTION:
Menopause is a natural process marking the end of the reproductive period and is accompanied by hormonal changes. These changes can significantly affect women's physical, emotional, mental, and social well-being. Symptoms experienced during and after the menopausal transition vary among individuals, and the severity of these symptoms may influence daily life activities. A woman's awareness of menopause and recognition of its symptoms play an important role in determining quality of life.

During menopause, the vascular and vasomotor systems, skeletal structure, and genitourinary system are commonly affected. Frequently reported symptoms include urinary incontinence, hot flashes, night sweats, vaginal problems, sleep disturbances, anxiety, irritability, and other physical and emotional changes. Genitourinary symptoms associated with hormonal changes may negatively affect women's quality of life and self-care abilities.

Urinary incontinence is a health problem that arises from dysfunction of the continence mechanism and has a profound impact on the quality of life of menopausal women. It is associated with various individual and environmental risk factors. Factors such as age, sociodemographic characteristics, reproductive history, chronic conditions, lifestyle factors, and obesity may contribute to the development of urinary incontinence during menopause.

As key members of the multidisciplinary healthcare team, nurses play an important role in identifying urinary incontinence, teaching and implementing conservative treatment methods, and providing counseling on preventive strategies. Management of urinary incontinence includes pharmacological and non-pharmacological treatments, behavioral approaches, and surgical interventions.

The Health Promotion Model focuses on understanding health-promoting behaviors and evaluating factors that influence these behaviors. The model emphasizes that health behaviors are shaped by individuals' past experiences and perceptions, and that thoughts guide actions. Its main concepts include the individual, environment, care, health, and illness.

Approaches based on health promotion models may strengthen women's ability to cope with symptoms related to urinary incontinence. In addition, the integration of internet-based tools and mobile applications into healthcare services plays an important role in supporting disease prevention, early detection, care, and treatment processes. These approaches facilitate access to healthcare services and enhance communication with healthcare professionals.

This study aims to evaluate the effects of education and counseling delivered through a mobile application based on a health promotion model on symptom severity, quality of life, and sleep quality in menopausal women with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

Outpatient admission to the Urology Clinic at Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital

Female, aged 40-65 years

Currently in menopause

Experiencing urinary incontinence

Literate (able to read and write)

Adequate comprehension and expression skills in Turkish

Ownership of an Android or iOS smartphone with internet access

Willingness to participate in the study

No diagnosed psychiatric disorders

Exclusion Criteria:

Withdrawal from the study by the participant

Not actively using the mobile application during the study period

Failure to complete required forms while using the mobile application

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopausal women
Enrollment: 82 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | up to 24 weeks
  The research data will be collected using a form developed by the researcher based on the literature, which includes participants' sociodemographic, obstetric, and gynecological information.
Urinary Incontinence Quality of Life Scale (I-QOL) | up to 24 weeks
  Developed by Wagner and Hu in 1998 to assess the quality of life of patients with urinary incontinence, the scale consists of 22 items and three subdimensions. Its validity and reliability in Turkish were established by Özer Doğan and colleagues. The subdimensions are: restriction of behaviors (items 1,2,3,4,10,11,13,20), psychosocial impact (items 5,6,7,9,15,16,17,21,22), and social isolation (items 8,12,14,18,19). All items are rated on a five-point Likert scale (1=very much, 2=quite a lot, 3=moderate, 4=a little, 5=none). The I-QOL and subscale scores are calculated by summing item scores and dividing by the number of items. To facilitate interpretation, the total score is converted to a scale from 0 (lowest quality of life) to 100 (highest quality of life). Higher scores indicate better quality of life.
Incontinence Severity Index (ISI) | up to 24 weeks
  Developed by Sandvik et al. in 1993 in Norway to evaluate the severity of urinary incontinence in women. The Turkish validity and reliability study was conducted by Hazar and Şirin in 2008. This simple, short, valid, and reliable scale is frequently recommended (level A) for severity assessment. The ISI consists of two questions, and the total score is obtained by multiplying the frequency of urine leakage by the amount leaked, ranging from 1 to 12. According to ISI scores, 1-2 points indicate mild; 3-6 moderate; 8-9 severe; and 12 very severe urinary incontinence. Mild incontinence typically refers to occasional drops of urine a few times a month, moderate to daily drops, and severe to at least once a week of large amounts of leakage. The Turkish validity and reliability study reported a Cronbach alpha of 0.67.
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | up to 24 weeks
  Developed by Avery et al. in 2004 to assess the prevalence, frequency, perceived cause, and impact of urinary incontinence on quality of life. The ICIQ consists of an unscored self-diagnostic item and three scored items. The Turkish validity and reliability study was conducted by Çetinel et al. in 2004. Cronbach's alpha was 0.71, with stability results of 0.98, 0.95, and 0.97 for questions 3, 4, and 5, respectively.
Pittsburgh Sleep Quality Index (PSQI) | up to 24 weeks
  Developed by Buysse et al. in 1989, with Turkish validity and reliability conducted by Ağargün et al. in 1996, reporting a Cronbach alpha of 0.79. PSQI is a self-report scale evaluating sleep quality and disturbances over the past month. The scale consists of 24 items in seven components: subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbances (component 5), use of sleep medication (component 6), and daytime dysfunction (component 7). The first 19 items are self-reported, while the last five are answered by a roommate or partner. Items are scored 0-3, with total scores ranging from 0 to 21. Higher scores indicate poorer sleep quality and greater disturbances. A total score above 5 indicates clinically poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No